CLINICAL TRIAL: NCT02674477
Title: Treatment Engagement With Technology-assisted Treatment
Acronym: TETAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00079236
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Results first posted 2019-07-19 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Alcoholism; Substance-related Disorders; Mentally Ill Chemical Abuse; Educational Technology
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Therapeutics

ARMS (2):
- Therapeutic Education System (TES) (Experimental): Participants will have the opportunity to use the TES program while hospitalized, at specific, monitored times, and can also use it when discharged by using participant's specific login information. Participants can use it as much or as little as participants like. Participants will continue with treatment as usual during and after hospitalization, as well.
  Interventions: Device: Therapeutic Education System (TES)
- Treatment as Usual (TAU) (Other): Standard treatment comprises a psychiatrist-led interdisciplinary team as well as face-to-face group counseling for substance use and skills for improving general mental health. There will be no change to the routine care (treatment at usual [TAU]) provided to patients on the service.
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Device: Therapeutic Education System (TES) — The TES program is made of modules about ways to prevent substance use, such as how to refuse drugs and alcohol, how to cope with thoughts about using, and how to make the best possible decisions for a person's mental health. Each module takes less than 30 minutes to complete. Modules may contain videos or other interactive media. At the end of each module, there are questions about the material.
  Arms: Therapeutic Education System (TES)
Other: Treatment as Usual (TAU) — Standard treatment comprises a psychiatrist-led interdisciplinary team as well as face-to-face group counseling for substance use and skills for improving general mental health. There will be no change to the routine care (treatment at usual [TAU]) provided to patients on the service.
  Arms: Treatment as Usual (TAU)

SUMMARY:
This research is being done to study whether using an Internet-based program, called the Therapeutic Education System (TES), would be helpful for the treatment of substance use and other psychiatric problems.

DETAILED DESCRIPTION:
TES has been shown to be helpful as substance abuse treatment in certain groups of people, mainly in the outpatient setting by using interactive modules for education. This study will expose some participants to this program while participants are hospitalized on an inpatient unit, and give the participants access to it after participants are discharged from the hospital. Those participants will still receive treatment as usual, as will the control group.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of drug or alcohol problem, plus another psychiatric problem, such as depression or anxiety
* drug or alcohol use in the last 30 days
* proficiency in English
* able to consent to study
* willing to engage in outpatient treatment
* willing to allow study team to contact outpatient providers

Exclusion Criteria:

* psychotic symptoms, such as hearing voices
* involuntary admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Strain, MD, Principal Investigator — Johns Hopkins University

REFERENCES:
- [Background] Chaple M, Sacks S, McKendrick K, Marsch LA, Belenko S, Leukefeld C, Prendergast M, French M. Feasibility of a computerized intervention for offenders with substance use disorders: a research note. J Exp Criminol. 2014;10(1):105-127. doi: 10.1007/s11292-013-9187-y. PMID 24634641
- [Background] Campbell AN, Nunes EV, Matthews AG, Stitzer M, Miele GM, Polsky D, Turrigiano E, Walters S, McClure EA, Kyle TL, Wahle A, Van Veldhuisen P, Goldman B, Babcock D, Stabile PQ, Winhusen T, Ghitza UE. Internet-delivered treatment for substance abuse: a multisite randomized controlled trial. Am J Psychiatry. 2014 Jun;171(6):683-90. doi: 10.1176/appi.ajp.2014.13081055. PMID 24700332
- [Derived] Hammond AS, Antoine DG, Stitzer ML, Strain EC. A Randomized and Controlled Acceptability Trial of an Internet-based Therapy among Inpatients with Co-occurring Substance Use and Other Psychiatric Disorders. J Dual Diagn. 2020 Oct;16(4):447-454. doi: 10.1080/15504263.2020.1794094. Epub 2020 Jul 23. PMID 32701419

RESULTS

PARTICIPANT FLOW:
Groups:
- Therapeutic Education System (TES): Participants will have the opportunity to use the TES program while hospitalized, at specific, monitored times, and can also use it when discharged by using their specific login information. They can use it as much or as little as they like. They will continue with treatment as usual during and after hospitalization, as well.
  Therapeutic Education System (TES): The TES program is made of modules about ways to prevent substance use, such as how to refuse drugs and alcohol, how to cope with thoughts about using, and how to make the best possible decisions for a person's mental health. Each module takes less than 30 minutes to complete. Modules may contain videos or other interactive media. At the end of each module, there are questions about the material.
- Treatment as Usual (TAU): Standard treatment comprises a psychiatrist-led interdisciplinary team as well as face-to-face group counseling for substance use and skills for improving general mental health. There will be no change to the routine care (treatment at usual [TAU]) provided to patients on the service.
  Treatment as Usual (TAU): Participants will received standard treatment during and after hospitalization.
Period: Overall Study
Arm/Group | Therapeutic Education System (TES) | Treatment as Usual (TAU)
Started | 48 | 47
Completed | 40 | 45
Not Completed | 8 | 2
Not completed — Protocol Violation | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Treatment as Usual (TAU): Participants will have the typical treatment during and after their hospitalizations, without additional intervention.
  Treatment as Usual (TAU): Participants will received standard treatment during and after hospitalization.
- Total: Total of all reporting groups
Arm/Group | Therapeutic Education System (TES) | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 48 | 47 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 47 | 95
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.5 (10.4) | 39.8 (8.1) | 39.01 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 33 | 31 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 48 | 44 | 92
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 16 | 18 | 34
  White | 32 | 27 | 59
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 47 | 95

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Treatment Based on Survey Questionnaire Completed by Participants
Description: The acceptability assessment asks about hospital satisfaction for both groups. The questionnaire is a series of questions on Qualtrics on a scale of 0-10. Higher scores signified a more positive response and a better outcome.
Time Frame: prior to discharge from the hospital up to 30 days
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Therapeutic Education System (TES) | Treatment as Usual (TAU)
Number analyzed (Participants) | 40 | 45
score on a scale | 8.78 (0.2) | 8.23 (0.3)

2. Secondary Outcome: Number of Participants Enrolled in Post-discharge Substance Abuse Treatment Appointments 30 Days After Hospital Discharge
Time Frame: 30 days after discharge from the hospital
Population: We only analyzed those who were referred to substance abuse treatment, and for whom we were able to receive the information from their treatment program
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Education System (TES) | Treatment as Usual (TAU)
Number analyzed (Participants) | 41 | 35
Participants | 23 | 19

3. Secondary Outcome: Number of Participants Enrolled in Post-discharge Treatment for Other Mental Health Appointments 30 Days After Hospital Discharge
Time Frame: 30 days after discharge from the hospital
Population: We only analyzed those who were referred to other mental health treatment, and for whom we were able to receive the information from their treatment program
Measure: Count of Participants; unit: Participants
Arm/Group | Therapeutic Education System (TES) | Treatment as Usual (TAU)
Number analyzed (Participants) | 36 | 39
Participants | 18 | 22

ADVERSE EVENTS:
Time Frame: 3 months after discharge from the hospital
Arm/Group | Therapeutic Education System (TES) | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/48 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-14): https://cdn.clinicaltrials.gov/large-docs/77/NCT02674477/Prot_SAP_000.pdf